CLINICAL TRIAL: NCT00249418
Title: Training Therapists to Administer Contingency Management-Patient Phase
Brief Title: Training Therapists to Administer Contingency Management-Patient Phase - 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-16855-3; R01DA016855 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Substance Abuse
Keywords: Contingency Management; Substance Abuse Treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management — Rewards (prizes) for abstinence

SUMMARY:
The purpose of this study is to train therapists to administer contingency management (CM). This project will train up to 42 community-based treatment providers about the rationale for and the specifics of administering CM. Initial training will occur in 2-day workshops, followed by weekly supervision in delivery of CM with test cases. We expect that the majority of therapists will achieve high levels of competence and adherence in administering CM treatment within 3-5 test cases, as measured by ratings of audiotapes. To examine the efficacy of CM, each therapist who achieves adherence and competence in delivering CM will administer standard treatment alone or standard treatment plus CM to substance-abusing outpatients. In the CM condition, patients will have the opportunity to win prizes for submission of negative samples, and the treatment will be in effect for 12 weeks. In total, up to 200 patients will be randomly assigned to one of the two conditions. A research evaluator will conduct follow-up assessments, scheduled for 3, 6 and 9 months after treatment initiation.

ELIGIBILITY:
Inclusion criteria:

* age 18 years or older
* meets DSM-IV criteria for cocaine abuse or dependence
* English speaking (est. >90% of patients)

For those in drug-free programs, they must have initiated treatment within the past week. For methadone patients, they must be stabilized on a dose of methadone, defined as being on the same dose for at least 30 days and not currently requesting or being considered for a dose modification. Methadone patients must also have submitted at least 30% cocaine positive urine samples in the past 3 months.

Exclusion criteria:

* acute uncontrolled psychiatric disorder (psychosis, suicidality) as determined by the SCID
* dementia (<23 on the Mini Mental State Exam; Folstein & Folstein, 1975)
* in recovery for pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and each follow-up
Retention | each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States